CLINICAL TRIAL: NCT04834362
Title: Efficacy and Safety of Human Insulin Versus Analog Insulin in Hospitalized Acute Stroke Patients With Hyperglycemia: a Randomized, Open-label, Single Center Trial
Brief Title: Insulin for Hyperglycemia in Stroke Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Neurosciences and Hospital, Dhaka (Other Government)
Responsible Party: Principal Investigator, Dr. Mashfiqul Hasan, Assistant Professor (Endocrinology), National Institute of Neurosciences and Hospital, Dhaka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108
Record Dates: First submitted 2021-03-26; First posted 2021-04-08 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Hyperglycemia; Stroke, Acute
Keywords: Hyperglycemia; Stroke; Human insulin; Analog insulin
MeSH Terms: conditions — Hyperglycemia; Stroke; Insulin Resistance | interventions — Insulin Aspart; Insulin Glargine; Insulin; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analog insulin arm (Experimental): Patients treated with insulin analog regimen will receive 50% of total daily dose as basal insulin glargine at the same time of day and 50% as insulin aspart given in 3 equally divided doses at 6 am, 12 pm and 6 pm.
  Interventions: Drug: Analog Insulin
- Human insulin arm (Active Comparator): Patients treated with human insulin regimen will receive 50% of total daily dose as NPH insulin at around 6 am and 6 pm, while the rest 50% regular human insulin three times a day in 3 equally divided doses at around 6 am, 12 pm and 6 pm
  Interventions: Drug: Human insulin

INTERVENTIONS:
Drug: Analog Insulin — For a patient who is known to have diabetes but were not getting insulin previously (or previous insulin dosage is not known), insulin therapy will be started at a total daily dose of 0.3-0.4 units/kg/day for an admission BG between 10-15 mmol/L or 0.5-0.6 units/kg/day for a BG >15 mmol/L. In previously insulin treated patients, ongoing total daily dose of insulin will be started. If there is history of poor glycemic control with ongoing insulin dose, then 10-20% increase of daily dose of insulin will be considered.
  For a patient who is not known to have diabetes, insulin therapy will be started if admission BG is >10 mmol/L in two or more occasions. A total daily dose of 0.3-0.4 units/kg/day will be started if admission BG is 10-15 mmol/L and 0.5-0.6 units/kg/day for a BG >15 mmol/L.
  Other Names: Insulin Aspart and Insulin Glargine
  Arms: Analog insulin arm
Drug: Human insulin — Patients treated with human insulin regimen will receive 50% of total daily dose as NPH insulin at around 6 am and 6 pm, while the rest 50% regular human insulin three times a day in 3 equally divided doses at around 6 am, 12 pm and 6 pm.
  Other Names: Regular insulin and NPH insulin
  Arms: Human insulin arm

SUMMARY:
Introduction: Glycemic control in acutely ill stroke patients with hyperglycemia is vital. Although insulin is the choice of anti-diabetic agent during acute stage, it is not clear which insulin regimen is better in terms of glycemic control and prevention of hypoglycemia in hospitalized acute stroke patients who are usually on small frequent nasogastric tube feeding. The present study aims to evaluate the efficacy and safety of human insulin (regular insulin and neutral protamine hagedorn, NPH insulin) to analog insulin (basal insulin glargine and rapid acting insulin aspart) in hospitalized acute stroke patients with hyperglycemia.

Justification: Analog insulins are developed by minor alteration of the amino acid chain which alters their pharmacokinetics and make them more physiological. However, these insulins are costly and are not widely available. Conventional human insulins are more commonly used in our country. Comparison of these two regimen is necessary in our own setting to optimize optimal glycemic management of hospitalized acute stroke patients.

Methodology: In this single-center, open-label, randomized trial, 100 patients with acute stroke and hyperglycemia (capillary blood glucose ≥10 mmol/L on 2 or more occasions) or history of type 2 DM admitted in the in-patient Department of Neurology, National Institute of Neurosciences (NINS) & Hospital will be randomly assigned to receive human insulin or modern insulin therapy in 1:1 ratio. The study will be carried out from February to June 2021. Blood glucose (BG) will be monitored by standardized glucometer thrice a day and insulin dose will be adjusted daily. The primary outcome of the study will be the differences in glycemic control between groups, as measured by mean daily BG concentration during the hospital stay. Secondary outcomes include differences between treatment groups in any of the following measures: number of hypoglycemic events (BG <3.9 mmol/L), total daily dose of insulin, length of hospital stay, hospital complications and mortality.

DETAILED DESCRIPTION:
METHODOLOGY:

Type of study: Single-center, open-label, randomized trial Place of Study: Department of Neurology, National Institute of Neurosciences & Hospital, Dhaka.

Study Period: February to June, 2021 Study population: Patients admitted in the Department of Neurology with acute stroke and hyperglycemia

Sample Size:

Sample size was calculated according to following formula for non-inferiority trial (17):

Here, N= sample size per group α= 0.05 β= 0.20 δ0= a clinically acceptable margin (assumed as 3 mmol/L of blood glucose) S2= Pooled standard deviation of both comparison group= 8 So,

As a result, 50 patients will be randomly assigned to two treatment groups (50 human insulin regimen, 50 analog insulin regimen).

Study Procedure Patients will be randomly assigned to receive either a human insulin regimen (starting with regular insulin three times a day with NPH insulin twice a day) or analog insulin regimen (basal insulin glargine once daily and insulin aspart three times a day) following a computer-generated randomization table. All oral antidiabetic drugs will be discontinued on admission.

For a patient who is known to have diabetes but were not getting insulin previously (or previous insulin dosage is not known), insulin therapy will be started at a total daily dose of 0.3-0.4 units/kg/day for an admission BG between 10-15 mmol/L or 0.5-0.6 units/kg/day for a BG >15 mmol/L. In previously insulin treated patients, ongoing total daily dose of insulin will be started. If there is history of poor glycemic control with ongoing insulin dose, then 10-20% increase of daily dose of insulin will be considered.

For a patient who is not known to have diabetes, insulin therapy will be started if admission BG is >10 mmol/L in two or more occasions. A total daily dose of 0.3-0.4 units/kg/day will be started if admission BG is 10-15 mmol/L and 0.5-0.6 units/kg/day for a BG >15 mmol/L.

Patients treated with human insulin regimen will receive 50% of total daily dose as NPH insulin at around 6 am and 6 pm, while the rest 50% regular human insulin three times a day in 3 equally divided doses at around 6 am, 12 pm and 6 pm.

Patients treated with modern insulin regimen will receive 50% of total daily dose as basal insulin glargine at the same time of day and 50% as insulin aspart given in 3 equally divided doses at 6 am, 12 pm and 6 pm.

In both groups, insulin dosage will be adjusted daily to a target fasting and premeal BG 7.8-10.0 mmol/L in the absence of hypoglycemia. Insulin dosage will be adjusted daily according to BG values. If the fasting and/or premeal BG is 10-15 mmol/L in the absence of hypoglycemia, the total daily dose will be increased by 10% every day. If the fasting and/or premeal BG is >15 mmol/L, the insulin daily dose will be increased by 20% every day. If a patient develops hypoglycemia (BG <3.9 mmol/L), the insulin daily dose will be decreased by 20%. Supplemental regular insulin will be given in addition to scheduled mealtime insulin for BG >10 mmol/L using a supplemental insulin protocol.

BG will be measured before each bolus insulin injection (at 6 am, 12 pm and 6 pm). Glycated hemoglobin (HbA1c) will be measured after hospital admission if not done within last three months. Except anti-diabetic treatment, other treatments will be continued as per the decisions of the treating physicians. If NG feeding is discontinued and patient is kept NPO, conventional group will receive neutralizing insulin with any dextrose containing fluid along with low dose NPH insulin, if needed. Modern insulin group will receive neutralizing insulin with any dextrose containing fluid with glargine insulin as before.

After recruitment, each recruited patient will be visited daily (even in holidays according to a predefined schedule) by one of the investigators and insulin dose will be adjusted according to glucose profile of previous day. Insulin injection and capillary blood glucose monitoring by glucometer will be done by trained nurses as part of their routine patient care. Doctors and nurses on duty will be provided with cell number of the investigators who will receive call on 24/7 basis for any emergency or uncertainty regarding management of hyperglycemia.

Hypoglycemia is regarded as the only short-term adverse event of insulin. As both treatment arms will use established and recognized insulin regimen, no compensation will be provided to the patient or his/her attendants in case of any adverse event. As most of the hospitalized patients have severe stroke with case fatality rate around 20%, death will not be regarded as parameter of primary treatment outcome.

During discharge, last in-hospital insulin dose will be continued with education to the caregiver regarding insulin injection and glucose monitoring technique. No follow up visit is included in the study.

Protocol deviation and protocol violation:

Deviation to protocol will be recorded and reported to ethical committee as soon as possible. Failure to obtain informed written consent, use of incorrect insulin regimen, not fulfilling inclusion and exclusion criteria will be regarded as protocol violation and will be reported to ethical committee immediately. In case of protocol violation, the data of related participant will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* • Patients admitted to adult neurology ward with acute stroke with

  * Patients having hyperglycemia (capillary blood glucose ≥10 mmol/L in 2 or more occasions or having history of treatment for DM)
  * Patients with age of 18-80 years of both sexes
  * Patients or their attendants giving consent to take part in the study

Exclusion Criteria:

* Patients with hyperglycemic emergencies (hyperglycemic hyperosmolar state or diabetic ketoacidosis)

  * Pregnant patients
  * Those not giving consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mashfiqul Hasan, MD, Principal Investigator — Assistant Professor (Endocrinology)
Locations (1):
- National Institute of Neurosciences and Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen R, Ovbiagele B, Feng W. Diabetes and Stroke: Epidemiology, Pathophysiology, Pharmaceuticals and Outcomes. Am J Med Sci. 2016 Apr;351(4):380-6. doi: 10.1016/j.amjms.2016.01.011. PMID 27079344
- [Background] Bellolio MF, Gilmore RM, Ganti L. Insulin for glycaemic control in acute ischaemic stroke. Cochrane Database Syst Rev. 2014 Jan 23;2014(1):CD005346. doi: 10.1002/14651858.CD005346.pub4. PMID 24453023
- [Result] Johnston KC, Bruno A, Pauls Q, Hall CE, Barrett KM, Barsan W, Fansler A, Van de Bruinhorst K, Janis S, Durkalski-Mauldin VL; Neurological Emergencies Treatment Trials Network and the SHINE Trial Investigators. Intensive vs Standard Treatment of Hyperglycemia and Functional Outcome in Patients With Acute Ischemic Stroke: The SHINE Randomized Clinical Trial. JAMA. 2019 Jul 23;322(4):326-335. doi: 10.1001/jama.2019.9346. PMID 31334795
- See also: Website of the study site — http://www.nins.gov.bd/nins/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants admitted to the study center with acute stroke were enrolled between April 2021 and June 2021. The first participant was enrolled on April 04, 2021 and the last participant was enrolled on June 14, 2021.
Pre-assignment Details: Of 452 enrolled participants, 105 met inclusion criteria and were randomized to treatment.
Groups:
- Analog Insulin Arm: Patients treated with insulin analog regimen will receive 50% of total daily dose as basal insulin glargine at the same time of day and 50% as insulin aspart given in 3 equally divided doses at 6 am, 12 pm and 6 pm.
  Analog Insulin: For a patient who is known to have diabetes but were not getting insulin previously (or previous insulin dosage is not known), insulin therapy will be started at a total daily dose of 0.3-0.4 units/kg/day for an admission BG between 10-15 mmol/L or 0.5-0.6 units/kg/day for a BG >15 mmol/L. In previously insulin treated patients, ongoing total daily dose of insulin will be started. If there is history of poor glycemic control with ongoing insulin dose, then 10-20% increase of daily dose of insulin will be considered.
  For a patient who is not known to have diabetes, insulin therapy will be started if admission BG is >10 mmol/L in two or more occasions. A total daily dose of 0.3-0.4 units/kg/day will be started if admission BG is 10-15 mmol/L and 0.5-0.6 units/kg/day for a BG >15 mmol/L.
Period: Overall Study
Arm/Group | Analog Insulin Arm | Human Insulin Arm
Started | 53 | 52
Completed | 52 | 50
Not Completed | 1 | 2
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Analog Insulin Arm | Human Insulin Arm | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (12.1) | 60.0 (11.4) | 59.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 23 | 25 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 52 | 50 | 102
Past history of Diabetes [Count of Participants; unit: Participants] | 41 | 45 | 86
NIHSS score [Mean (Standard Deviation); unit: units on a scale] — National Institutes of Health Stroke Scale (NIHSS) The maximum possible score is 42, with the minimum score being a 0. Higher score indicates more severity of stroke.
  units on a scale | 16 (6) | 15 (7) | 15 (6)
GCS score [Mean (Standard Deviation); unit: units on a scale] — Glasgow coma scale (GCS) score measures the consciousness. Maximum score 15, minimum 3. Lower score indicates lower consciousness.
  units on a scale | 11 (3) | 11 (3) | 11 (3)
Systolic blood pressure [Mean (Standard Deviation); unit: mm of Hg] | 146 (20) | 147 (24) | 146 (22)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm of Hg] | 91 (13) | 89 (13) | 90 (13)
HbA1c [Mean (Standard Deviation); unit: %] | 9.9 (2.8) | 10.2 (2.2) | 10.0 (2.5)
S. Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.13 (0.53) | 1.19 (0.61) | 1.15 (0.56)
Feeding pattern on admission [Count of Participants; unit: Participants]
  Nasogastric tube feeding | 26 | 34 | 60
  Oral feeding | 14 | 11 | 25
  Nothing per oral | 12 | 5 | 17
Feeding pattern during outcome [Count of Participants; unit: Participants]
  Nasogastric tube feeding | 24 | 26 | 50
  Oral feeding | 20 | 18 | 38
  Nothing per oral | 8 | 6 | 14
Use of steroids [Count of Participants; unit: Participants] | 20 | 20 | 40
Stroke type [Count of Participants; unit: Participants]
  Ischemic | 28 | 24 | 52
  Hemorrhagic | 24 | 26 | 50
NIHSS category [Count of Participants; unit: Participants] — National Institutes of Health Stroke Scale (NIHSS) The maximum possible score is 42, with the minimum score being a 0. Higher score indicates more severity of stroke.
  Score 1-4: Mild Score 5-15: Moderate Score 16-20: Severe Score 21-42: Very severe
  Participants
    Score 1-4 | 3 | 4 | 7
    Score 5-15 | 14 | 19 | 33
    Score 16-20 | 27 | 19 | 46
    Score 21-42 | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Differences in glycemic control between groups, as measured by mean blood glucose concentration
Time Frame: During the hospital stay assessed up to 10 days
Population: According to inclusion and exclusion criteria 105 patients were randomized in the study. Of them 102 were analyzed at the end of trial. 52 received analog insulin and 50 received human insulin.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Analog Insulin Arm | Human Insulin Arm
Number analyzed (Participants) | 52 | 50
mmol/L | 10.7 (2.9) | 10.9 (3.0)
Statistical Analysis 1: Comparison: Analog Insulin Arm vs Human Insulin Arm; Test type: Other; p = 0.677, t-test, 2 sided

2. Secondary Outcome: Total Daily Dose of Insulin
Description: Total daily dose of insulin is calculated according to total basal insulin dose plus total bolus insulin dose divided by days of treatment
Time Frame: During the hospital stay assessed up to 10 days
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Analog Insulin Arm | Human Insulin Arm
Number analyzed (Participants) | 52 | 50
Units/day | 22.3 (8.8) | 26.7 (13.3)
Statistical Analysis 1: Comparison: Analog Insulin Arm vs Human Insulin Arm; Test type: Other; p = 0.053, t-test, 2 sided

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay of the study participants
Time Frame: During the hospital stay assessed up to 10 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Analog Insulin Arm | Human Insulin Arm
Number analyzed (Participants) | 52 | 50
Days | 4.7 (2.5) | 4.8 (2.3)
Statistical Analysis 1: Comparison: Analog Insulin Arm vs Human Insulin Arm; Test type: Other; p = 0.918, t-test, 2 sided

4. Secondary Outcome: Mortality
Description: In-hospital mortality of the study participants
Time Frame: During the hospital stay assessed up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Analog Insulin Arm | Human Insulin Arm
Number analyzed (Participants) | 52 | 50
Participants | 15 | 16
Statistical Analysis 1: Comparison: Analog Insulin Arm vs Human Insulin Arm; Test type: Other; p = 0.729, Chi-squared

ADVERSE EVENTS:
Time Frame: During the period of hospitalization, up to 10 days.
Arm/Group | Analog Insulin Arm | Human Insulin Arm
All-Cause Mortality (participants affected / at risk) | 15/52 | 16/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 9/52 | 10/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Analog Insulin Arm (N=52) | Human Insulin Arm (N=50)
Hypoglycemia (Investigations) | 9 (10) | 10 (15) — Hypoglycemic events in the study participants, defined as blood glucose <3.9 mmol/L

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04834362/Prot_SAP_001.pdf